CLINICAL TRIAL: NCT02801071
Title: "Treatment With L-citrulline in Patients With Post-polio Syndrome - a Randomized Double Blind Placebo Controlled Study"
Brief Title: L-Citrulline in Patients With Post-Polio Syndrome
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Dirk Fischer (Other)
Responsible Party: Sponsor-Investigator, Dirk Fischer, Prof. Dr. med., University Hospital, Basel, Switzerland
Organization: University Hospital, Basel, Switzerland (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PPS
Record Dates: First submitted 2016-06-06; First posted 2016-06-15 (Estimated); Last update posted 2019-01-23 (Actual); Status verified 2019-01

CONDITIONS: Post-Polio Syndrome
Keywords: Post-Polio Syndrome; PPS
MeSH Terms: conditions — Postpoliomyelitis Syndrome

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- L-citrulline (Experimental): 15 g L-citrulline p.o. per day (3x 5g) for 24 weeks
  Interventions: Drug: 15g L-citrulline daily p.o.
- Placebo (Placebo Comparator): L-citrulline Placebo 3 times daily p.o. for 24 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: 15g L-citrulline daily p.o.
  Arms: L-citrulline
Drug: Placebo
  Arms: Placebo

SUMMARY:
The purpose of the study is to show that the intake of L-citrulline improves muscle function in patients with Post-Polio Syndrome (PPS).

DETAILED DESCRIPTION:
This is a single center, randomized, double-blind, placebo controlled study. The study medication consists of L-citrulline, respectively placebo given orally; 5 g L-citrulline or placebo will be given three times daily. The duration of the study is 48 weeks and comprehends one screening and four study visits.

Additionally, in order to investigate whether PPS is associated with an atrophy of spinal cord gray and potentially also white matter as well as motor cortex atrophy, it is planned to offer all trial participants an additional optional spinal cord/brain MRI investigation and a MRI at week 48 and a follow-up one year later together with a clinical and physiotherapy assessment during extension phase. We don't expect Citrulline to affect the spinal cord gray or white and gray matter.

ELIGIBILITY:
Inclusion Criteria:

* Prior paralytic poliomyelitis with evidence of motor neuron loss
* A period of partial or complete functional recovery after acute paralytic Poliomyelitis
* Slowly progressive and persistent new muscle weakness or decreased endurance, with or without generalized fatigue, muscle atrophy, or muscle and joint pain. Symptoms that persist for at least a year
* Exclusion of other neuromuscular, medical and skeletal abnormalities as causes of symptoms
* Patients older than 18 years at time of Screening
* ambulant
* ability to walk 150m in the 6 min. Walking distance (6MWD)
* females of childbearing potential willing to use contraceptive during the study

Exclusion Criteria:

* Previous (3 months or less) or concomitant participation in any other therapeutic trial
* Use of L-citrulline or L-arginine within the last 3 months
* Known individual hypersensitivity to L-citrulline
* Known or suspected malignancy
* Other chronic disease or clinical relevant limitation of renal, liver, heart function according to discretion of investigator
* Pregnant or breast-feeding women
* Severe renal failure (calculated glomerular filtration rate (GFR) < 30 ml/min)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2016-06-14 (Actual); Primary Completion 2017-08-15 (Actual); Study Completion 2018-10-05 (Actual)

PRIMARY OUTCOMES:
Mean change of 6 Minute Walking Distance(6MWD) | Baseline to week 48

SECONDARY OUTCOMES:
Mean change of motor function measure (MFM) total score | Baseline to week 48
Change of quantitative muscle MRI (IDEAL-CPMG with T₂ and lipid quantitation and dynamic 31P-MR spectroscopy) | Baseline to week 48
Change of serum concentrations for markers of muscle necrosis | Baseline to week 48
Change of serum concentrations for markers of oxidative stress | Baseline to week 48
Change of serum concentrations for markers of nitrosative stress | Baseline to week 48
Change of serum concentrations for markers of mitochondrial related genes | Baseline to week 48

OTHER OUTCOMES:
Change of disease severity measured by questionnaires | Baseline to week 48
  Mean change of disease severity as assessed by a combination of the Self-Reported Impairments in Persons With Late Effects of Polio Rating Scale (SIPP-RS), the Inclusion Body Myositis Functional Rating Scale (IBM-FRS) and the World Health Organization Quality Of Life (WHOQOL-BREF)
Changes in Spinal cord MRI from week 48 to week 96 | week 48 to week 96
  1. Determination of the degree of spinal cord gray and white matter atrophy in PPS patients in comparison to healthy controls and its relationship to physical disability (QMT).
  2. Determination of the degree of motor cortex atrophy in PPS patients compared to healthy controls and its association with spinal cord gray and white matter atrophy in PPS patients.
  3. Determination of the association between spinal cord gray matter atrophy and microstructural alterations as assessed by diffusion tensor imaging.
  4. Test the suitability of the applied, optimized imaging and post-processing methods for longitudinal data.
Changes in brain MRI from week 48 to week 96 | week 48 to week 96
  1. Determination of the degree of spinal cord gray and white matter atrophy in PPS patients in comparison to healthy controls and its relationship to physical disability (QMT).
  2. Determination of the degree of motor cortex atrophy in PPS patients compared to healthy controls and its association with spinal cord gray and white matter atrophy in PPS patients.
  3. Determination of the association between spinal cord gray matter atrophy and microstructural alterations as assessed by diffusion tensor imaging.
  4. Test the suitability of the applied, optimized imaging and post-processing methods for longitudinal data.

CONTACTS AND LOCATIONS:
Overall Officials: Dirk Fischer, Prof., Principal Investigator — University Children's Hospital Basel
Locations (1):
- University of Basel, Children's Hospital, Basel, Switzerland

REFERENCES:
- [Derived] Gocheva V, Hafner P, Orsini AL, Schmidt S, Schaedelin S, Rueedi N, Rubino-Nacht D, Weber P, Fischer D. Health-related quality of life, self-reported impairments and activities of daily living in relation to muscle function in post-polio syndrome. J Patient Rep Outcomes. 2020 Jul 16;4(1):59. doi: 10.1186/s41687-020-00226-5. PMID 32676980
- [Derived] Schmidt S, Gocheva V, Zumbrunn T, Rubino-Nacht D, Bonati U, Fischer D, Hafner P. Treatment with L-citrulline in patients with post-polio syndrome: study protocol for a single-center, randomised, placebo-controlled, double-blind trial. Trials. 2017 Mar 9;18(1):116. doi: 10.1186/s13063-017-1829-3. PMID 28274276